CLINICAL TRIAL: NCT00125736
Title: A Double-blind, Comparative Study in Patients With Gastric Ulcer to Evaluate the Efficacy of Combination Use of E0671 and Rabeprazole Sodium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E0671-J081-291
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2010-01

CONDITIONS: Stomach Ulcer
MeSH Terms: conditions — Stomach Ulcer | interventions — Rabeprazole

ARMS (2):
- E0671 combination group (Experimental)
  Interventions: Drug: E0671; Drug: rabeprazole sodium
- placebo combination group (Placebo Comparator)
  Interventions: Drug: rabeprazole sodium; Drug: E0671 placebo

INTERVENTIONS:
Drug: E0671 — One 50 mg capsule is orally administered three times daily (150 mg/day)
  Arms: E0671 combination group
Drug: rabeprazole sodium — One 10mg tablet is administered orally each day
Drug: E0671 placebo — One 50 mg capsule is orally administered three times daily (150 mg/day)
  Arms: placebo combination group

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of combination use of E0671 and Rabeprazole Sodium in patients with gastric ulcer.

DETAILED DESCRIPTION:
The efficacy and safety of E0671 in combination with Rabeprazole Sodium (i.e., 10 mg/day of rabeprazole sodium and 150 mg/day of E0671) will be investigated in patients with gastric ulcer in a multicenter, randomized, double-blind, parallel-group comparative study using a placebo control group (10 mg/day of rabeprazole sodium and placebo for E0671).

ELIGIBILITY:
Inclusion criteria:

1. Patients with gastric ulcer (A1-and A2-stage)
2. Patients with gastric ulcer who meet all of the following items. Gender and treatment class (in-patient or out-patient) are not asked.

   * Patients with endoscopically diagnosed A1- or A2-stage ulcer (by Sakita/Miwa classification).
   * Patients who are not younger than 20 years of age at the time of obtaining informed consent.
   * Patients who meet any of the following conditions:

     * H. pylori-negative
     * H. pylori-positive and not requiring eradication therapy
     * H. pylori-positive and unsuccessful eradication
3. Patients who are given a full explanation about the study objective and design, and able to give prior consent for study participation.

Exclusion criteria:

1. Patients with a complication of duodenal ulcer (excluding cicatrix).
2. Patients with reflux esophagitis
3. Patients with acute gastric mucosal lesions (AGML).
4. Patients with NSAID-induced ulcer.
5. Patients with linear ulcer.
6. Patients with ulcer injured by endoscopy.
7. Patients who underwent gastrectomy or vagal nerve resection.
8. Patients who are not applied to pharmacotherapy, i.e., perforation, pyloric stenosis, major bleeding (exposed blood vessels in the base of ulcer), etc.
9. Patients receiving proton pump inhibitor (PPI) and/or teprenone preparation(s) within 1 week prior to the study administration.
10. Patients with serious cardiovascular diseases (e.g., angina pectoris, heart failure, acute myocardial ischemia, severe tachyarrhythmia), serious hematological disorders (e.g., aplastic anemia), serious renal disorders (e.g., acute, chronic renal failure), serious hepatic disorders (e.g., cirrhosis, severe hepatitis), serious pancreatic disorders (e.g., severe pancreatitis), serious psychoneuroses (e.g., schizophrenia, alcoholic dependency, drug dependency, severe depression), or cancer.
11. Patients with a current or a history of drug allergy to teprenone preparation(s).
12. Patients with a current or a history of drug allergy to PPI.
13. Patients requiring antacid(s) containing digoxin or aluminum hydroxide/magnesium hydroxide that are suspected to exert drug interaction with rabeprazole sodium.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2005-08-01 (Actual); Primary Completion 2007-04-19 (Actual); Study Completion 2007-04-19 (Actual)

PRIMARY OUTCOMES:
Ratio of S2-stage transition at 8 weeks after the study administration. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshihisa Arai, Study Director — GI Group. Post-Marketing Clinical Research Dept., Clinical Research Center
Locations (43):
- Japan (43):
  - Kariya, Aichi-ken
  - Nagoya, Aichi-ken
  - Seto, Aichi-ken
  - Toyoake, Aichi-ken
  - Toyohashi, Aichi-ken
  - Akita, Akira
  - Urayasu, Chiba
  - Niihama, Ehime
  - Chikushino-shi, Fukoka
  - Fukoka, Fukoka
  - Kurume, Fukoka
  - Oumuta, Fukoka
  - Tagawa, Fukoka
  - Sabae, Fukui
  - Hashima, Gifu
  - Asahikawa, Hokkaido
  - Sapporo, Hokkaido
  - Miki, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Kumamotoi, Kumamoto
  - Sendai, Miyagi
  - Kashihara, Nara
  - Nigata, Niigata
  - Yufu, Oita Prefecture
  - Ikeda, Osaka
  - Izumisano, Osaka
  - Kadoma, Osaka
  - Takatsuki, Osaka
  - Hasuda, Saitama
  - Kitaadachi-gun, Saitama
  - Matsue, Shimane
  - Hamamatsu, Shizouka
  - Minato-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjyuku-ku, Tokyo
  - Shimonoseki, Yamaguchi
  - Gifu
  - Hiroshima
  - Kouchi
  - Kyoto
  - Nara
  - Ōita
  - Saga